CLINICAL TRIAL: NCT05771311
Title: Potassium Tetanyl Phosphate Laser vs Pulsed Dye Laser for Treating Port-Wine Stains - A Prospective, Split-Side Study
Brief Title: KTP Laser vs Pulsed Dye Laser for Port-Wine Stains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-21
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Titanyle Phosphate (KTP) Laser (Active Comparator): split-side, 1 - 5 sessions at intervals of 6 - 8 weeks
  Interventions: Device: KTP
- Pulsed Dye Laser (Active Comparator): split-side, 1 - 5 sessions at intervals of 6 - 8 weeks
  Interventions: Device: PDL

INTERVENTIONS:
Device: KTP — split-side, 1 -5 sessions at intervals of 6 - 8 weeks
  Arms: Potassium Titanyle Phosphate (KTP) Laser
Device: PDL — split-side, 1 -5 sessions at intervals of 6 - 8 weeks
  Arms: Pulsed Dye Laser

SUMMARY:
To compare the efficacy and safety of 532nm KTP laser and 585 nm pulsed dye laser for treating port-wine stains.

DETAILED DESCRIPTION:
Nevus flammeus is a vascular, primarily capillary malformation visible from birth on. In rare cases, it may also affect venous and/or arterial vascular systems of the skin or other organs [1]. It occurs in 0.3%-0.5% of the population [1], i.e. in about 3-4 out of 1000 newborns, and is thus the most frequent vascular malformation in children. The cause is a permanent dilatation of the capillary vessels, which is caused by a lack of sympathetic nerve fibers or a lower density of the same.

First-line therapy of port-wine stains consists of laser treatment with the long-pulsed dye laser [2] with a wavelength of 595nm. Treatment must be performed at least 10 times at intervals of about 8 weeks and leads to lightening and reduction of lesions. In recent years, problems have often arisen in care of port-wine stain patients because dye lasers often failed due to the instability of technology, resulting in treatment delays. Novel long-pulsed KTP lasers may be a sufficient alternative to pulsed dye lasers in treatment of port-wine stains.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and older
* Good general health, no relevant previous diseases
* Presence of one or more port-wine stains
* Cognitive ability and willingness to give consent (Informed Consent)

Exclusion Criteria:

* Age < 18 years
* Pregnant and breastfeeding women
* Significant open wounds or lesions in the region to be treated
* Missing consent and/or data protection declarations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Erythema | at follow-up visit 6 weeks after last treatment session
  assessment scale 1 - 7 (normal skin - dark purple) evaluated by physician and blinded investigator
area reduction | at follow-up visit 6 weeks after last treatment session
  measurement using photo documentation

SECONDARY OUTCOMES:
patient satisfaction | at follow-up visit 6 weeks after last treatment session
  assessment scale 1 - 6 (very - not at all) evaluated by subjects

CONTACTS AND LOCATIONS:
Overall Officials: L Nguyen, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Laser Department, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen JK, Ghasri P, Aguilar G, van Drooge AM, Wolkerstorfer A, Kelly KM, Heger M. An overview of clinical and experimental treatment modalities for port wine stains. J Am Acad Dermatol. 2012 Aug;67(2):289-304. doi: 10.1016/j.jaad.2011.11.938. Epub 2012 Feb 3. PMID 22305042
- [Background] Updyke KM, Khachemoune A. Port-Wine Stains: A Focused Review on Their Management. J Drugs Dermatol. 2017 Nov 1;16(11):1145-1151. PMID 29141064